CLINICAL TRIAL: NCT03559400
Title: A Pilot Masked, Randomized Controlled Trial Evaluating Locally-applied Gentamicin Versus Saline in Open Tibia Fractures
Brief Title: Pilot RCT Local Gentamicin for Open Tibial Fractures in Tanzania
Acronym: pGO-Tibia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Muhimbili Orthopaedic Institute (Other); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17-23950; K23AR079044 (NIH)
Record Dates: First submitted 2018-06-06; First posted 2018-06-18 (Actual); Results first posted 2023-12-22 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Open Tibia Fracture

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients will receive gentamicin in saline solution or placebo saline injection while under anesthesia during the index surgery. Only the local research pharmacist, the UCSF clinical trial manager, and the DSMC will be unmasked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- gentamicin injection at fracture site (Experimental): Subjects with an open tibia fracture who receive gentamicin in saline solution administered after closure at the time of initial debridement.
  Interventions: Drug: local gentamicin injection
- placebo saline injection at fracture site (Placebo Comparator): Subjects with an open tibia fracture who receive placebo saline solution administered after closure at the time of initial debridement.
  Interventions: Drug: placebo saline injection

INTERVENTIONS:
Drug: local gentamicin injection — Treatment includes debridement and administration of the local antibiotic which will consist of 80mg of liquid gentamicin diluted in 40mL normal saline injected after inserting a 22 gauge needle down to bone after wound closure. The injection will continue until either all 40cc are injected or there is fluid extravasation from the wound.
  Arms: gentamicin injection at fracture site
Drug: placebo saline injection — Treatment includes debridement and administration of the local antibiotic which will consist of 40mL normal saline injected after inserting a 22 gauge needle down to bone after wound closure. The injection will continue until either all 40cc are injected or there is fluid extravasation from the wound.
  Arms: placebo saline injection at fracture site

SUMMARY:
Local application of antibiotics directly to the traumatic wound is a promising strategy for the prevention of infection after open tibia fractures, which are a significant source of disease burden globally, particularly in low-income countries. This pilot study aims to assess feasibility of a randomized controlled trial to measure the effect of locally applied gentamicin on risk of infection for open tibial fractures in Tanzania. If proven effective, local gentamicin would be a highly cost-effective strategy to reduce complications and disability from open tibial fractures that could impact care in both high- and low-income countries.

DETAILED DESCRIPTION:
This pilot study is being conducted in Dar es Salaam, Tanzania to assess the feasibility of a masked, placebo-controlled, randomized trial to compare local gentamicin injection to saline injection in open tibial shaft fractures. The study will enroll patients within 1 week of injury. The active or placebo agent will be administered during the initial surgical debridement based on a web-based randomization tool. Patients will be followed for 1 year after surgery to assess for the occurrence of fracture-related infection (FRI), a consensus definition of infection after open fracture or insertion of internal fixation to treat fracture. Additional clinical and economic endpoints will also be measured.

Depending on the outcome of the feasibility study, we may undertake a definitive trial to test the effectiveness of local gentamicin to prevent FRI. If proven effective, local gentamicin would impact the clinical care of open fracture patients both in Tanzania and likely in high-income settings as well. These data will also deepen the understanding of the clinical and economic impact of FRI in open fracture populations.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients age 18 or older
2. Diagnosis of an acute open tibial shaft fracture meeting the following criteria:

   1. AO/OTA Type 42
   2. Primarily closable wound
   3. Type I, II, or IIIA Gustilo- Anderson (GA) Classification

Exclusion Criteria:

1. Time from injury to presentation > 48 hours
2. Time from injury to surgery >7 days
3. History of Aminoglycoside allergy
4. GA IIIB or IIIC open fractures
5. Bilateral open tibial fractures
6. Severe brain (GCS<12) or spinal cord injury
7. Severe vascular injury
8. Sustained severe burns (>10% total body surface area (TBSA) or >5% TBSA with full thickness or circumferential injury)
9. Pathologic fracture
10. History of active limb infection, ipsilaterally

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-11-19 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Shearer, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- Muhimbili Orthopaedic Institute, Dar es Salaam, Tanzania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] von Kaeppler EP, Donnelley C, Ali SH, Roberts HJ, Ibrahim JM, Wu HH, Eliezer EN, Porco TC, Haonga BT, Morshed S, Shearer DW. A study protocol for a Pilot Masked, Randomized Controlled Trial Evaluating Locally-applied Gentamicin versus Saline in Open Tibia Fractures (pGO-Tibia) in Dar es Salaam, Tanzania. Pilot Feasibility Stud. 2021 Feb 10;7(1):47. doi: 10.1186/s40814-021-00766-7. PMID 33568230

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gentamicin Injection at Fracture Site | Placebo Saline Injection at Fracture Site
Started | 45 | 55
Completed | 36 | 46
Not Completed | 9 | 9
Not completed — Lost to Follow-up | 9 | 7
Not completed — Death | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gentamicin Injection at Fracture Site | Placebo Saline Injection at Fracture Site | Total
Number analyzed (Participants) | 45 | 55 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.9 (14) | 32.5 (11) | 33.6 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 8 | 20
  Male | 33 | 47 | 80
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Tanzania | 45 | 55 | 100
Mechanism of Injury [Count of Participants; unit: Participants]
  Road Traffic Injury | 37 | 47 | 84
  Fall | 2 | 3 | 5
  Crush Injury | 2 | 3 | 5
  Gunshot | 2 | 0 | 2
  Other | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Rate of Enrollment
Description: The number of participants enrolled in the clinical trial per month will be measured to assess feasibility of the definitive clinical trial.
Time Frame: Baseline
Population: For pilot trial feasibility aims, the outcomes are presented for all trial participants rather than by arm to match the a priori feasibility targets for the definitive trial.
Measure: Mean (Full Range); unit: Participants enrolled per month
Groups:
- Overall Enrollment: Subjects who were enrolled and randomized to either local gentamicin or placebo saline injection.
Arm/Group | Overall Enrollment
Number analyzed (Participants) | 100
Participants enrolled per month | 12.5 [7 to 17]

2. Primary Outcome: Rate of Retention
Description: The percentage of patients completing 1 year follow up relative to the total number of participants
Time Frame: 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Enrollment
Number analyzed (Participants) | 100
Participants | 84

3. Primary Outcome: Occurrence of Fracture-related Infection (FRI)
Description: The primary outcome for the definitive trial is occurrence of fracture-related infection (FRI), a binary variable. Any of the four following diagnostic criteria are confirmatory for FRI:
  1. fistula, sinus or wound breakdown
  2. purulent drainage from the wound or presence of pus during surgery
  3. phenotypically indistinguishable pathogens identified by culture from at least two separate deep tissue/implant specimens
  4. presence of microorganisms in deep tissue taken during an operative intervention, as seen on histopathological examination.
  All primary events will be reviewed by a masked adjudication committee comprised of 3 non-treating fellowship-trained orthopaedic trauma surgeons.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Gentamicin Injection at Fracture Site | Placebo Saline Injection at Fracture Site
Number analyzed (Participants) | 37 | 46
Participants | 9 | 7

4. Secondary Outcome: Euro-Qol 5 Dimensions (EQ-5D)
Description: EuroQol-5 Dimensions (EQ-5D) measures general health status in five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The raw score will be translated to a utility score ranging from 0 (death or no health) to 1 (perfect health) on a continuous scale using health-state valuations from Zimbabwe.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: units on a scale from 0 to 1
Arm/Group | Gentamicin Injection at Fracture Site | Placebo Saline Injection at Fracture Site
Number analyzed (Participants) | 45 | 55
units on a scale from 0 to 1 | 0.950 (0.101) | 0.938 (0.195)

5. Secondary Outcome: Modified Radiographic Union Scale for Tibial Fractures (mRUST) Score
Description: Radiographic healing as measured by the modified Radiographic Union Scale for Tibial fractures (mRUST). mRUST scores each cortex on an AP and lateral radiograph from a score of 1 (no callus) to 4 (remodeled, fracture not visible). Thus, mRUST ranges from 4 (worst healing score) to 16 (best healing score).
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: score on a scale from 4-16
Arm/Group | Gentamicin Injection at Fracture Site | Placebo Saline Injection at Fracture Site
Number analyzed (Participants) | 45 | 55
score on a scale from 4-16 | 11.9 (2.9) | 12.0 (3.1)

6. Secondary Outcome: Function Index for Trauma (FIX-IT) Score
Description: Clinical healing of the fracture will be assessed using the Function index for trauma (FIX-IT) score, which evaluates weight bearing and pain in patients with lower extremity fractures. The FIX-IT score is a clinical outcomes assessment measure ranging from 0 to 12 points in two domains: the ability to bear weight (maximum 6 points) and pain at the fracture site (maximum 6 points). The maximum score of 12 indicates the highest level of function.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Gentamicin Injection at Fracture Site | Placebo Saline Injection at Fracture Site
Number analyzed (Participants) | 45 | 55
score on a scale | 10.9 (2.7) | 11.2 (2.5)

7. Secondary Outcome: Occurrence of Nonunion
Description: Nonunion is a binary variable defined by the following criteria:
  1. any unplanned reoperation for promotion of bone healing; OR
  2. mRUST<=10 AND either: FIX-IT score <=11 at 12-month follow-up OR recommendation by treating surgeon for nonunion repair surgery
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Gentamicin Injection at Fracture Site | Placebo Saline Injection at Fracture Site
Number analyzed (Participants) | 45 | 55
Participants | 7 | 6

8. Secondary Outcome: Occurrence of Fracture-related Reoperation
Description: This binary variable includes reoperation for infection, wound healing, or fracture union, and excludes the removal of implants for prominence/irritation.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Gentamicin Injection at Fracture Site | Placebo Saline Injection at Fracture Site
Number analyzed (Participants) | 45 | 55
Participants | 3 | 1

9. Other Pre Specified Outcome: Direct Medical Costs
Description: Direct medical costs of treatment (continuous), including medications, personnel, and supplies will be measured for both the intervention and control groups.
Time Frame: 1 year
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Indirect Medical Costs
Description: Indirect (time) costs, such as lost productivity, will be measured using the Work Productivity and Activity Impairment questionaire (WPAI)
Time Frame: 1 year
Reporting Status: Not Posted

11. Other Pre Specified Outcome: C-Reactive Protein Level
Description: C-Reactive protein (CRP) is a known inflammatory marker which may show signs of early infection. The value will be measured in all patients and reported at 6 weeks post-surgery.
Time Frame: 6 weeks
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Microbiology of FRI
Description: For cases undergoing reoperation for which deep tissue cultures are taken, the frequency of each bacterial species will be reported as a percentage of total FRI for both treatment groups.
Time Frame: 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 Year
Description: Definitions consistent with clinicaltrials.gov.
  All participants were screened for kidney injury using pre and post-operative creatinine levels. Hearing loss and urinary problems were assessed using a standard questionnaire at each follow up.
Arm/Group | Gentamicin Injection at Fracture Site | Placebo Saline Injection at Fracture Site
All-Cause Mortality (participants affected / at risk) | 0/45 | 2/55
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/55
Other Adverse Events (participants affected / at risk) | 5/45 | 5/55
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gentamicin Injection at Fracture Site (N=45) | Placebo Saline Injection at Fracture Site (N=55)
Acute Kidney Injury (Renal and urinary disorders) | 5 (5) | 4 (4) — Mild to moderate acute kidney injury, defined as a 0.3-1.0 above baseline creatinine
Hearing impairment (Ear and labyrinth disorders) | 0 (0) | 1 (1) — Hearing impairment reported on screening questionairre

LIMITATIONS AND CAVEATS:
This feasibility study was predictably underpowered to detect differences in fracture-related infection and other clinically important secondary outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-05-18): https://cdn.clinicaltrials.gov/large-docs/00/NCT03559400/Prot_SAP_000.pdf
  • Informed Consent Form (2021-05-27): https://cdn.clinicaltrials.gov/large-docs/00/NCT03559400/ICF_001.pdf